CLINICAL TRIAL: NCT07082153
Title: A Prospective, Multicenter Clinical trIal in Evaluating the Safety and Efficacy of the Coronary Sinus Balloon Pump for the First-In-Man Use in STEMI Patients
Brief Title: The First-In-Man Use of Coronary Sinus Balloon Pump in STEMI Patients Treated by Primary PCI
Acronym: REVIVE-FIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort Rhythm MedTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REVIVE-FIM
Record Dates: First submitted 2025-05-12; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: STEMI
Keywords: STEMI; the coronary sinus balloon pump
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The coronary sinus balloon pump (Experimental): Subjects in experimental group will be treated with the coronary sinus balloon pump manufactured by Shanghai Microport Rhythm Co. Ltd.
  Interventions: Device: the coronary sinus balloon pump

INTERVENTIONS:
Device: the coronary sinus balloon pump — The coronary sinus balloon pump comprises a coronary sinus balloon pump catheter system and a coronary sinus balloon pump therapeutic device. This product is indicated for the treatment of ST-segment elevation myocardial infarction (STEMI) with or without coronary microvascular dysfunction (CMD), by intermittently occluding coronary sinus blood flow during percutaneous coronary intervention (PCI) procedures to reduce myocardial infarction size.

SUMMARY:
This is a prospective, multicenter clinical investigation aiming to evaluate the safety and efficacy of the coronary sinus balloon pump in its first application in patients with acute ST-segment elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
This is a prospective, multicenter clinical investigation to evaluate the safety and efficacy of the coronary sinus balloon pump in its first application in patients with acute ST-segment elevation myocardial infarction (STEMI).

The target population for this clinical study consists exclusively of patients diagnosed with acute ST-segment elevation myocardial infarction (STEMI) who require emergency percutaneous coronary intervention (PCI) treatment.

The clinical outcome data collected will be based on the site's standards of care for acute STEMI. Examinations include but are not limited to physical assessments, cardiac markers, ECG, laboratory results, x-rays, angiograms, cMRI, and echocardiography.

Endpoint data will be collected at multiple follow-up intervals: during CSBP therapy, immediately following device explantation, at 5 days and 30 days post-procedure, and subsequently at 4-month, 6-month, and 12-month follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

Clinical inclusion criteria：

1. Subjects aged ≥18 and ≤80 years with clinically confirmed ST-segment elevation myocardial infarction (STEMI).
2. Left Ventricular Dysfunction: Left ventricular ejection fraction (LVEF) ≤50% assessed by pre-PCI echocardiography or left ventriculography.
3. Ischemic Symptoms: Presence of myocardial infarction symptoms consistent with ischemic timing (e.g., persistent chest pain, with or without dyspnea, nausea/vomiting, diaphoresis, syncope), with symptom onset between 6 and 24 hours prior to enrollment.
4. Electrocardiographic Evidence:

   * Acute anterior wall myocardial infarction confirmed by 12-lead ECG, demonstrating ST-segment elevation ≥1 mm (0.1 mV) in ≥2 contiguous precordial leads.
   * For leads V2 or V3:

   Men: ST-segment elevation ≥2 mm (0.2 mV) Women: ST-segment elevation ≥1.5 mm (0.15 mV).
5. PCI Eligibility: Candidate for primary percutaneous coronary intervention (PCI).
6. Subjects who can understand the purpose of the trial, voluntarily participate and acknowledge the risks and benefits described in the informed consent document by signing the informed consent form, and can conscientiously complete clinical follow-up as required

Angiography Inclusion Criteria:

1. Target Lesion Location: Located in the proximal or mid segment of the Left Anterior Descending artery (LAD).
2. Pre-PCI TIMI Flow: TIMI flow grade 0 or 1 in the target vessel prior to percutaneous coronary intervention (PCI).

Exclusion Criteria:

1. Presence of implants or foreign bodies within the coronary sinus.
2. Target lesion involving the left main coronary artery or ≥50% stenosis in the left main coronary artery.
3. Known hypersensitivity to medications or devices required during PCI or the investigational device (including but not limited to: rapamycin, polyurethane in dual antiplatelet therapy, PET, or stainless steel).
4. Pericardial effusion (moderate or larger volume), cardiac tamponade, hemodynamically significant left/right shunts, or severe valvular heart disease.
5. Intracardiac thrombus detected by echocardiography within 30 days prior to enrollment.
6. History of acute myocardial infarction (AMI) or documented hospitalization for Q-wave infarction.
7. History of cerebral infarction, intracranial hemorrhage, transient ischemic attack (TIA), or reversible ischemic neurologic deficit within the past 6 months, or permanent neurological deficits.
8. Hemoglobin <90 g/L, platelet count <80×10⁹/L, history of bleeding disorders/coagulopathy, or refusal to accept blood transfusion.
9. Requiring circulatory support or assisted ventilation therapy.
10. Cardiac arrest or cardiopulmonary resuscitation (CPR) >5 minutes during pre-procedural baseline or intra-procedural period.
11. Unsuitable femoral or jugular venous access.
12. Contraindications to cardiac magnetic resonance imaging (CMR), including claustrophobia, CMR-incompatible implants/foreign bodies, or gadolinium contrast allergy/intolerance.
13. Prior coronary artery bypass grafting (CABG).
14. Visible collateral circulation formation distal to the target lesion in the target vessel.
15. Current participation in another investigational drug/device trial (prior to primary endpoint completion) or planned enrollment in another trial within 12 months post-procedure.
16. Severe renal dysfunction (eGFR <30 mL/min/1.73m² by MDRD equation*) or ongoing hemodialysis.
17. Active malignancy treatment within the past 12 months.
18. Chronic obstructive pulmonary disease (COPD) requiring home oxygen therapy or chronic steroid therapy.
19. Impaired consciousness during PCI, cardiogenic shock (persistent SBP ≤90 mmHg despite conservative therapy), or pulmonary edema (peripheral SpO₂ <90% with rales).
20. Any vascular PCI performed within 7 days prior to hospitalization.
21. Fibrinolytic therapy administered within 24 hours prior to hospitalization.
22. Non-target lesions requiring treatment during index PCI or within 1 week post-procedure (excluding LAD and its branches).
23. Pregnancy, lactation, or female subjects planning pregnancy within 1 year post-procedure unable to complete follow-up.
24. Poor protocol compliance per investigator's judgment, or subjects deemed ineligible due to other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-12 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-03 (Estimated)

PRIMARY OUTCOMES:
Device-related procedural complication rate | 24 hours, 30 days post-procedure
  Device-related procedural complication rate [24 hours, 30 days post-procedure]:
  Complications include:
  * Access site complications: BARC type 3-5 bleeding; infection requiring oral/intravenous antibiotics; or access site complications requiring surgical intervention
  * Coronary sinus dissection or perforation requiring interventional/surgical treatment
  * Pericardial effusion or cardiac tamponade requiring interventional/surgical treatment
  * Thrombosis or embolism
  * Stroke (Note: CEC adjudication required to determine device-relatedness)

SECONDARY OUTCOMES:
MACCE (Major Adverse Cardiac and Cerebrovascular Events) | 5 days, 30 days, 4 months, 6 months, 12 months post-procedure
  MACCE (Major Adverse Cardiac and Cerebrovascular Events) [5 days, 30 days, 4 months, 6 months, 12 months post-procedure]:
  * Cardiac death
  * Hospitalization for heart failure
  * New-onset heart failure or worsening of pre-existing heart failure
  * Ventricular tachycardia/fibrillation requiring cardioversion/defibrillation
  * Myocardial infarction (MI)
  * Target vessel revascularization (TVR)
  * Stent thrombosis
  * Major bleeding (BARC type 3-5)
  * Stroke

OTHER OUTCOMES:
All-cause mortality rate (cardiac, vascular, non-vascular) | 5 days, 30 days, 4 months, 6 months, 12 months post-procedure
Heart failure hospitalization rate | 30 days, 4 months, 6 months, 12 months post-procedure
New-onset/worsening heart failure rate | 30 days, 4 months, 6 months, 12 months post-procedure
MI incidence | 5 days, 30 days, 4 months, 6 months, 12 months post-procedure
Revascularization rate | 5 days, 30 days, 4 months, 6 months, 12 months post-procedure
  Revascularization rate (target lesion, target vessel, any coronary)
Stent thrombosis rate | 5 days, 30 days, 4 months, 6 months, 12 months post-procedure
Major bleeding rate (BARC type 3-5) | 5 days, 30 days, 4 months, 6 months, 12 months post-procedure
  Based on the Bleeding Academic Research Consortium (BARC) Scale, type 5 is more serious.
Stroke incidence | 5 days, 30 days, 4 months, 6 months, 12 months post-procedure
Adverse event (AE)/Serious adverse event (SAE) rate | Periprocedural, 5 days, 30 days, 4 months, 6 months, 12 months post-procedure
Device deficiency rate | Periprocedural, 5 days, 30 days, 4 months, 6 months, 12 months post-procedure
Device success rate | Periprocedural
  Successful device delivery to the coronary sinus, deployment, and completion of therapy
Procedure success rate | Periprocedural
  PCI success without CSBP-related adverse events (based on device success)
Coronary sinus pressure | intra-procedure
MRI measurement of infarct size | 5 days, 4 months post-procedure
Angina severity | 5 days, 30 days, 4 months, 6 months, 12 months post-procedure
  Angina severity (classified according to the Canadian Cardiovascular Society Classification of Angina Pectoris) is assessed by the level of physical activity that triggers the chest pain. And the lower the level that triggers the chest pain, the more serious angina.
Changes in quality of life | 5 days, 30 days, 4 months, 6 months, 12 months post-procedure
  Changes in quality of life measured by EQ-5D (assessed by the following five dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression) (scale of 0-100: higher score better)
Assessment of left ventricular function | 5 days, 4 months post-procedure
  Left ventricular function assessed by echocardiography